CLINICAL TRIAL: NCT04230343
Title: Limits of the Social Benefit Motive Among High-risk Patients: a Field Experiment on Influenza
Brief Title: Limits of the Social Benefit Motive Among High-risk Patients: a Field Experiment on Influenza Vaccination Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Burcu Isler, Principal investigator, SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 855 - 21/10/2016
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Influenza Vaccine; Behavioral Intervention; Self-benefit; Social-benefit
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-benefit arm (Experimental)
  Interventions: Behavioral: Self-benefit message
- Social-benefit arm (Active Comparator)
  Interventions: Behavioral: Other-benefit message

INTERVENTIONS:
Behavioral: Self-benefit message — A pamphlet consisting of a short text and an abstract figure. The top half of the pamphlet described the official criteria for qualifying to be in the risk group. Bottom half indicated that one can gain immunity against influenza by getting the vaccine and included a figure of one smiley face.
  Arms: Self-benefit arm
Behavioral: Other-benefit message — A pamphlet consisting of a short text and an abstract figure. The top half of the pamphlet described the official criteria for qualifying to be in the risk group. Bottom half indicated that one can gain immunity against influenza by getting the vaccine, and gaining immunity would lower the chances of transmitting the disease to others. The figure included one smiley face surrounded by three other smiley faces.
  Arms: Social-benefit arm

SUMMARY:
Influenza vaccine uptake remains low worldwide, inflicting substantial costs to public health and health systems. Messages promoting social welfare have been shown to increase vaccination intentions, and it has been recommended that health professionals communicate the socially beneficial aspects of vaccination. This study aims to provide the first test whether this prosocial vaccination hypothesis applies to the actual vaccination behaviour of high-risk patients by comparing the effects of two motivational messages for promoting vaccination at a tertiary care public hospital in Istanbul, Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at medical departments of the hospital who are on the day of discharge

Exclusion Criteria:

* Egg ellergy
* Previous allergic reaction to influenza vaccine
* Pregnancy
* Cognitive disability

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2016-11-13 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
Vaccine uptake following the introduction of the pamphlet | On the same day, upto 24 hours
  Difference in the number of patients in each arm who agree to receive influenza vaccine following the introduction of the pamphlet. The first half of the pamphlet contains information about the the influenza vaccine and the risk groups who are vulnerable to influenza-associated serious diseases. The second half introduces the self-benefit message. And the final part asks if the participant wants to receive the influenza vaccine now.

SECONDARY OUTCOMES:
Vaccine uptake in high and low risk group patients following the introduction of the pamphlet | On the same day, upto 24 hours
  Vaccine uptake in high and low risk group patients. The first half of the pamphlet contains information about the the influenza vaccine and the risk groups who are vulnerable to influenza-associated serious diseases. The second half introduces the social-benefit message. And the final part asks if the participant wants to receive the influenza vaccine now.

CONTACTS AND LOCATIONS:
Locations (1):
- SB Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isler O, Isler B, Kopsacheilis O, Ferguson E. Limits of the social-benefit motive among high-risk patients: a field experiment on influenza vaccination behaviour. BMC Public Health. 2020 Feb 17;20(1):240. doi: 10.1186/s12889-020-8246-3. PMID 32066407